CLINICAL TRIAL: NCT06123390
Title: Cluster-Randomized Trial of the Implementation of the Responses to Illness Severity Quantification System (RISQ) in Children With Acute Malnutrition Six to Fifty-nine Months of Age in Ngouri, Chad
Brief Title: Evaluating RISQ System Implementation in Acutely Malnourished Children in Chad (CRIMSON)
Acronym: CRIMSON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Alliance for International Medical Action (Other); University of N'Djaména, Chad (Unknown)
Responsible Party: Principal Investigator, Christopher Parshuram, Staff Physician, Paediatric Intensive Care Unit, Department of Critical Care Medicine, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1000080735
Record Dates: First submitted 2023-10-26; First posted 2023-11-08 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Severe Acute Malnutrition
Keywords: decision support; mortality; illness severity; risk score
MeSH Terms: conditions — Severe Acute Malnutrition | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: In this study we are evaluating usual care (Arm 1) vs. the Responses to Illness Severity Quantification (Arm 2) in children children aged 6 to 59 months who are enrolled in the OptiMA nutrition program in Chad.
  Community health centres will be the randomized clusters.
Who Masked: Outcomes Assessor
Masking Description: The participants and care providers will know which arm of the study they are part of, as the randomization occurs at the facility level. Only the statistician will be blinded to the arms at the time of analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): The 17 health centres randomized to "Usual Care" will provide care as per OptiMA program.
- Intervention Arm (Experimental): The 17 health centres randomized to the intervention arm will provide care as per OptiMA program with the addition of the RISQ System decision support.
  Interventions: Other: The Responses to Illness Severity Quantification (RISQ) System

INTERVENTIONS:
Other: The Responses to Illness Severity Quantification (RISQ) System — The RISQ System involves: [1] the RISQ score: calculated routinely using the [2] documentation record and linked to [3] score-matched recommendations. Introduction into clinical care is supported by [4] the RISQ System implementation package. During the 2 month prior to implementation, front-line staff in the intervention arm will be trained on and will practice the use of the RISQ System .
  Arms: Intervention Arm

SUMMARY:
The purpose of this study is to evaluate the effect of the Responses to Illness Severity Quantification (RISQ) system implementation on mortality and processes of care in a nutritional program treating children 6 to 59 months of age with acute malnutrition in Ngouri, Chad.

DETAILED DESCRIPTION:
The CRIMSON Study is a 12-month cluster randomized trial that will evaluate the effect of implementing the RISQ system compared with usual care on all-cause mortality, in children with acute malnutrition aged 6 to 59 months enrolled in the OptiMA nutrition program in Chad.

The intervention is the RISQ System and the clusters are the individual health centres that are randomized with a ratio of 1:1, RISQ System: Usual care. The 12 month intervention period will begin following a run in phase in which sites randomized to intervention will introduce and establish the new practices and in which sites randomized to usual care will continue to provide usual care.

The RISQ system is a scientifically developed clinical decision support tool that consists of: [1] the RISQ score; [2] documentation form; [3] score-matched recommendations and [4] an implementation package. The RISQ score, developed through our prospective observational study in Maiduguri Nigeria ((NCT04582773) ranges from 0 to 26 (high scores indicating greatest severity of illness). In the development dataset, the mean RISQ score on admission was 3.6 in hospital survivors and 7.3 for children dying <48hr of admission. RISQ scores <24hr before death had Area Under the Receiver Operating Characteristics Curve (AUROC) of 0.93. The RISQ score performed similarly well in children independent of their clinical conditions as a diagnosis-independent measure of severity of illness. Additionally, through a study of 903 hospitalized children with Severe Acute Malnutrition (SAM), the RISQ score could discriminate between points of escalation or de-escalation of care and can reflect illness severity in children throughout hospitalization. The documentation form provides visual representation of the sub-scores of each RISQ score items and guidance for score calculation. The score-matched recommendations of the RISQ system that are linked to the RISQ scores are derived from an expert panel of clinicians, with over 100 years of collective experience caring for acutely malnourished children, and provide guidance about intensity of care. This includes the frequency of observation, consideration of secondary review, inpatient admission, and transfer into / out of inpatient care areas where more intensive treatments are provided.The implementation package consists of theoretical and practical training modules including specific 'train the trainers' sessions for key personal involved in the implementing programs.

The CRIMSON study is nested within the existing framework of the OptiMA nutritional program and observational study conducted by the Alliance for International Medical Action (ALIMA). The program involves health centres within Ngouri, a sub-prefecture of the Lake Region in Chad (and surrounding area) plus an inpatient unit at the Ngouri District Hospital providing care for children with acute malnutrition. Inclusion criteria for the OptiMA program are based on mid-upper arm circumference (MUAC) of <125mm and/or bilateral pitting oedema. Usual care in the OptiMA program is as follows: nutritional treatment to participants consists of Ready-to-use-Therapeutic Food (RUTF) adjusted based on their MUAC value throughout the duration of their care. Management of the children with acute illnesses follows the established approach for management of children with severe acute malnutrition using the World Health Organization (WHO) "danger signs" and Integrated Management of Childhood Illness (IMCI) algorithms to guide admission to hospital. Additionally, as part of the OptiMA program in Ngouri, pulse oximeters have been introduced in all health centres and inpatient care unit, following training by ALIMA. Included in the routine visits of the program is the measurement and documentation of each of the 7 RISQ score items [heart rate, respiratory rate, respiratory effort, oxygen saturation, temperature, level of consciousness and oxygen use (oxygen is currently only available in the inpatient care)] by nurses.

The investigators anticipate that implementation of the RISQ system in a nutrition treatment program will improve sensitivity and specificity of clinical evaluation in determining which children require hospitalization, and what level of medical care within the in-patient unit is appropriate and in turn potentially reduce mortality.

ELIGIBILITY:
Inclusion Criteria:

Children:

1. age: 6 to 59 months at enrolment on the day of their admission/re-admission to the OptiMA program
2. written consent to participate

Front line staff providing care to patients enrolled in the Optima program:

[1] Registered Nurses [2] Medical Doctors

Exclusion Criteria:

Children:

1. Children allergic to milk, peanuts and/or ready-to-use therapeutic food (RUTF)
2. Children not residing in one of the study areas.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20000 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality. | 12 months
  Mortality over the period beginning at admission to the program and ending at either program discharge or to a maximum of 60 days after study enrolment. Program discharge will be one of: [1] medical/anthropometric criteria or [2] defaulting from the program.
  Defaulting from the program is defined as children who do not attend the weekly clinic visits for 3 consecutive weeks.

SECONDARY OUTCOMES:
Timing of inpatient mortality | Duration of hospitalization in days up to 60 days
  Timing will be defined as [a] within 48 hours of hospital admission and [b] timing of death after admission to hospital
Timing of outpatient mortality | Duration of program inclusion in days up to 60 days
  Timing will be defined as [a] within 48 hours of being seen by health-care team [b] timing of death after being seen by outpatient health-care team
Therapeutic intensity | First 24 hours from admission to hospital
  To be measured by location on admission to inpatient care (Intensive Care Unit/Phase1/Phase2)
Efficiency of inpatient care | Duration of hospitalization in days up to 60 days
  Efficiency measured by length of inpatient stay (whole or part days)
Workload | Month 1 and month 12
  Frontline staff perception of workload measured through questionnaires using a 5 point scale
Knowledge | Month 1 and month 12
  Frontline staff knowledge of assessment skills measured through questionnaire using a 5 point scale
Fidelity of RISQ Implementation | 12 months
  Number of measured vital signs performed on individual patient at health centre visit with corresponding disposition in program, recorded in 10 randomly selected patients/week/health centre
Acceptability | Month 1 and month 12
  Acceptability of the RISQ System by front-line staff evaluated through a questionnaire using a 5 point scale

OTHER OUTCOMES:
Lived experience of RISQ System implementation | one time at end of 12 month implementation period
  Lived experiences measured by open ended questions about strengths/weaknesses of RISQ System implementation added to frontline staff perception questionnaire at end of intervention period
comparison of automated versus manual measurements of vital signs (Respiratory rate in breaths/min) | During run-in phase prior to implementation of intervention, on average 2 months
  Comparison determined by agreement between the two different methods for respiratory rate measurement
comparison of automated versus manual measurements of vital signs (Temperature in degrees Celsius) | During run-in phase prior to implementation of intervention, on average 2 months
  Comparison determined by agreement between the two different methods for temperature measurement
Comparison of RISQ scores among children with different clinical conditions in inpatient care | Duration of hospitalization in days up to 60 days
  Differences in RISQ scores among children with different clinical diagnoses a) on admission to inpatient care; b) throughout inpatient care; and c) at exit from inpatient care

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Parshuram, MD, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Ngouri, Ngouri, Chad

IPD SHARING:
Plan to Share IPD: No
On reasonable request - after publication of the study and with permission of parties attached to the study, and after Research Ethics Board review and approval.

REFERENCES:
- [Background] Dale NM, Ashir GM, Maryah LB, Shepherd S, Tomlinson G, Briend A, Zlotkin S, Parshuram C. Development and an initial validation of the Responses to Illness Severity Quantification (RISQ) score for severely malnourished children. Acta Paediatr. 2022 Sep;111(9):1752-1763. doi: 10.1111/apa.16410. Epub 2022 Jun 3. PMID 35582782
- [Background] Dale NM, Ashir GM, Maryah LB, Shepherd S, Tomlinson G, Briend A, Zlotkin S, Parshuram CS. Evaluating the Validity of the Responses to Illness Severity Quantification Score to Discriminate Illness Severity and Level of Care Transitions in Hospitalized Children with Severe Acute Malnutrition. J Pediatr. 2023 Nov;262:113609. doi: 10.1016/j.jpeds.2023.113609. Epub 2023 Jul 5. PMID 37419241
- [Derived] Dale NM, Hagre YD, Shepherd S, Tomlinson G, Zlotkin S, Ngaradoum M, Bechir M, Madjissem M, Tehoua C, Parshuram C. Cluster-randomized trial of the implementation of the Responses to Illness Severity Quantification (RISQ) system in children with acute malnutrition 6 to 59 months of age in Ngouri, Chad: the CRIMSON trial protocol. Trials. 2025 Jun 3;26(1):188. doi: 10.1186/s13063-025-08871-1. PMID 40462129
- See also: World Health Organization. Guideline: Updates on the Management of Severe Acute Malnutrition in Infants and Children [Internet]. 2013. — http://apps.who.int/iris/bitstream/10665/95584/1/9789241506328_eng.pdf
- See also: World Health Organization. Pocket Book of Hospital Care for Children: Guidelines for the Management of Common Childhood Illnesses, 2013. — http://www.ncbi.nlm.nih.gov/books/NBK154447/
- See also: World Health Organization. Handbook IMCI: Integrated Management of Childhood Illness [Internet]. 2005. — http://apps.who.int/iris/bitstream/10665/42939/1/9241546441.pdf
- See also: Exploratory meeting to review new evidence for Integrated Management of Childhood Illness (IMCI) danger signs — https://www.who.int/publications-detail-redirect/WHO-MCA-19.02